CLINICAL TRIAL: NCT03343938
Title: Comparative Study Between Two Systems of Gamete and Embryo Handling: Closed Environment Versus Open System
Brief Title: Evaluation of a Closed Assisted Reproductive Technology (ART) Station Versus an Open Flow Cabinet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1605-SEV-036-NP
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: ART
Keywords: Group embryo culture; Low oxygen tension; Closed station; Embryo handling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed Station (Experimental): Embryo handling is performed inside a closed station with a controlled environment: 6% CO2 and 37 degrees.
  Interventions: Other: Embryo handling in a closed station
- Open flow cabinet (No Intervention): Embryo handling is performed inside a conventional open flow cabinet without a controlled environment.

INTERVENTIONS:
Other: Embryo handling in a closed station — Embryo handling is performed inside a closed station with a controlled environment: 6% CO2 and 37 degrees.
  Arms: Closed Station

SUMMARY:
There is not yet a standardized system of human embryonic culture in vitro. In addition, technical improvements continually appear. The investigators recently carried out a study in which it shows that the grouped embryo culture at low oxygen tension (5% O2) in a benchtop incubator shows better success rates than individual culture at atmospheric oxygen tension (20% O2) in a conventional incubator. For these reasons, the investigators have decided to continue this research line to evaluate the efficacy of a new ART station with a closed environment in comparison of an open flow cabinet. This new system keeps a controled environment maintaining a carbon dioxide (CO2) concentration of 6% and a temperature of 37 degrees. A prospective randomized study will be carried out in which the manipulation of the gametes and pre-embryos of the patients will be carried out in open laminar flow cabinets or in a closed station that maintain the CO2 and temperature conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signing a written consent to participate in the study.
* Blastocyst transfer:
* Patients using their own oocytes under 40 years.
* Patients using donated oocytes.

Exclusion Criteria:

* Preimplantation genetic screening patients.
* Severe male factor (spermatozoa of testicular or epididymal origin, patients with cryptozoospermia and patients with retrograde ejaculation)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Embryo quality | Through study completion, an average of two years
  Rate of viable embryos = Transferred and Frozen embryos / Total number of embryos obtained

SECONDARY OUTCOMES:
Live birth rate per first embryo transfer | Through study completion, an average of two years
  Total number of live births over the total of recruited patients (taking into account only the first cycle)
Cumulative live birth rate | Through study completion, an average of two years
  Total number of live births over the total of recruited patients (taking into account fresh and cryopreserved cycles)
Implantation rate | Through study completion, an average of two years
  Total of implanted embryos / total of transferred embryos
Live birth rate of the first cycle per transferred embryo | Through study completion, an average of two years
  Total number of live births over the total of transferred embryo

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No